CLINICAL TRIAL: NCT02889068
Title: Targeted Next Generation Sequencing and Intellectual Disability
Acronym: NGS-DI
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2014/NGSDI-BONNET/NK
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen DNA from blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intellectual disability
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
The purpose is to determine the benefit of next generation sequencing (NGS) targeted on genes involved in intellectual disability for etiologic diagnosis of intellectual disabilities. In other words, it concerns the number of patients whose etiologic diagnosis will be established with NGS and could not with common techniques. Actually, the molecular etiology of intellectual disability is crucial to calculate the risk of recurrence and allows the perinatal diagnosis to these families.

Secondary purposes are:

1. To determine the place of NGS in the strategy of etiologic diagnosis of intellectual disability, to determine the order of analyses performed for a patient with intellectual disability without clinical signs.
2. To evaluate the number of variants with unknown significance and thus non-usable for genetic counselling without supplementary analysis.
3. To determine the number of samples that can be at most pooled keeping a good efficacy of capture and results with suitable read depth
4. To determine the possibility of detecting copy number variations (CNVs) in genes of interest with NGS
5. To establish genotype/phenotype correlations for each gene for which a mutation has been identified
6. To optimize the software pipelining for a rapid analysis for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe intellectual disability
* Availability of patient and parent DNA
* No etiologic diagnosis with standard approaches: negative fragile X, normal pangenomic 180K and 1M array-CGH
* Informed consent of person having parental authority

Exclusion Criteria:

* Non availability of parent DNA
* Patient lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe to moderate intellectual disability, with syndrome or not.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with certain etiologic diagnosis established with NGS | day 0

SECONDARY OUTCOMES:
Percentage of patients with etiologic diagnosis established with NGS or with other techniques (array-CGH) | day 0
Obtained read depth according to number of pooled samples | day 0
Percentage of patients with variant with unknown significance, needing supplementary analyses to prove its involvement in intellectual disability | day 0
CNVs detected with NGS or array-CGH (reference technique for CNV detection). | day 0
Clinical phenotype for each gene for which a causal mutation is identified by NGS | day 0
Time of analysis of NGS raw data | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Céline BONNET, Principal Investigator — CHRU de Nancy Laboratoire de Génétique Hôpitaux de Brabois
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No